CLINICAL TRIAL: NCT02142790
Title: Weekly and Every 3 Week Administration of Paclitaxel Liposome Injection in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Luye Sike Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY-TM-LPS-2014-02
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- paclitaxel liposome injection weekly (Experimental): paclitaxel liposome injection 100mg/m2 administered by intravenous on day1 and day8 of a 21-day cycle for at least 4cycles or till progression or intolerable
  Interventions: Drug: paclitaxel liposome injection
- paclitaxel liposome injection every 3 weeks (Experimental): paclitaxel liposome injection 175mg/m2 administered by intravenous on day1 of a 21-day cycle for at least 4cycles or till progression or intolerable
  Interventions: Drug: paclitaxel liposome injection

INTERVENTIONS:
Drug: paclitaxel liposome injection
  Other Names: LIPUSU

SUMMARY:
This is a open-label study in patients with metastatic breast cancer to evaluate the antitumor activity and safety of weekly dose-dense paclitaxel liposome injection compared to 3-weekly regimen.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male >18 years of age and < 70years of age, If female of childbearing potential, pregnancy test is negative before first dose of study drug and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study
* Stage IV disease
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Suitable for the treatment with paclitaxel as single agent regimen (first line or prior first line chemotherapy including adriamycin is allowed, If a taxane was part of the adjuvant regimen, at least one year should have transpired since completion of taxane regimen and if Her2+ patient, Herceptin therapy will be allowed.
* Patient has the following values at Baseline: Absolute neutrophil count ≥ 1.5 x 10^9cells/L; platelets ≥ 100 x 10^9 cells/L; hemoglobin ≥ 10 g/dL. Aspartate transaminase (AST or SGOT), alanine aminotransferase (ALT or SGPT) ≤ 2.5x upper limit of normal range (ULN); total bilirubin ≤ 1.5ULN; creatinine ≤ 1.5 mg/dL.
* Informed consent has been obtained.

Exclusion Criteria:

* Parenchymal brain metastases.
* History of other malignancy within the last 3 years
* New York Heart Association (NYHA) Grade 2 or greater congestive heart failure,history of myocardial infarction or unstable angina or new occured angina within 6 months prior to study enrollment.
* Concurrent other anticancer therapy.
* History of serious organic disorders (including active infection or Cardiovascular disease), serious hepatic disease, serious blood coagulation diseases, cachexia
* Sensory neuropathy of > Grade 1 at baseline.
* Patients with prior hypersensitivity to paclitaxel
* Pregnant or nursing women
* enrolled in a different clinical study
* No psychiatric illness and other situations that would limit compliance of study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 24 months

SECONDARY OUTCOMES:
Overall Response Rate | 24 months
Clinical Benefit Rate | 24 months
Adverse Events | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China